CLINICAL TRIAL: NCT04603105
Title: Clinical Characterisation Protocol for Severe Emerging Infections in the UK (CCP-UK) - a Prospective Companion Study for Patients With Cancer and COVID-19
Brief Title: CCP Cancer UK Companion Study
Status: Active, not recruiting | Type: Observational
Sponsor: The Clatterbridge Cancer Centre NHS Foundation Trust (Other)
Collaborators: University of Edinburgh (Other); University of Oxford (Other); University of Liverpool (Other)
Responsible Party: Sponsor
Other Study IDs: C1147
Record Dates: First submitted 2020-10-09; First posted 2020-10-26 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Cancer; Covid19
MeSH Terms: conditions — Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Study Cohort: Patients will be recruited from the main study after being determined to having COVID-19 and Cancer

SUMMARY:
Currently, there is extremely limited information regarding the risks posed by SARS-CoV-2 to patients with cancer. This study aims to understand the presentation, management and outcomes of patients with cancer. The influence of cancer type and treatment will be explored as well as comparing cancer patients with non-cancer patients. This dataset, on robust analysis, will provide valuable information that would educate as well as help inform practice for future possible outbreaks. The information may also inform the development of guidelines with regard to the care and management of cancer patients with viruses such as COVID19 and similar infectious diseases. Cancer is immunosuppressive, the nature of the immunosuppression seems to be influenced by the microbiota, and in addition pulmonary infections

DETAILED DESCRIPTION:
In December 2019 the first pneumonia cases of unknown origin were identified in Wuhan, the capital city of Hubei province. High-throughput sequencing revealed the pathogen to be a novel enveloped RNA betacoronavirus. Initially named 2019 novel coronavirus (2019-nCoV) it was subsequently renamed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) (2). Transmission of SARS-CoV-2 is via respiratory droplets and direct contact, and infection results in coronavirus disease (COVID-19). The World Health Organization (WHO) has recently declared the SARS-CoV-2 outbreak a public health emergency of international concern on 30th January 2020, and a global pandemic on 11th March 2020.

The clinical characteristics of COVID-19 are typically fever, dry cough and fatigue, sometimes accompanied by sore throat, chest discomfort and difficulty breathing. However, a wide range of other symptoms are possible, including gastrointestinal symptoms such as nausea, vomiting, loss of appetite, abdominal pain and diarrhoea. Loss of taste and smell have also been described.

Individuals with malignant disease are more prone to respiratory viruses than individuals without cancer as a result of immunosuppression caused by either the underlying disease process or systemic anti-cancer therapy. The death rate from influenza in patients with solid organ tumours is much higher than expected for the background population, even allowing for likely ascertainment bias. This is reflected in individuals with cancer being recommended to receive the seasonal flu vaccination. Certain groups of cancer patients are even more prone to infection. For example, patients with haematological malignancy undergoing bone marrow transplantation have significant mortality even with rhinovirus, which can double the transplant related mortality. There is currently no prospective robust data regarding the presentation, management and outcome of patients with COVID-19 with cancer who are immunocompromised as result of either the disease or treatment. Furthermore, it is not clear if the immunosuppressive effects of systemic anti-cancer therapy such as chemotherapy are the same across all cancer types and the possible risks entailed by targeted therapies and immunotherapy. Currently, cancer patients on treatment are considered at high risk group of possible severe infection with SARS-CoV-2 and measures such as self-isolation are being recommended to mitigate the risks of such patients being infected. However, information to inform this decision, and whether any specific sub-groups of patients are at particular risk is lacking. These data are vital to inform policy on cancer treatments as patients may be potentially exposed to SARS-CoV-2 for a long time to come. Furthermore, given patients with cancer are often immunosuppressed and this may alter the clinical presentation as well as clinical course and outcomes. Different tumour types may also have implications for SARS-CoV-2 exposure, for example patients with lung cancer may be more susceptible, and require different pathways to ensure care can be delivered safely. This protocol aims to describe the presentation, management and outcomes of patients with solid and haematological malignancies with COVID-19 and compared to non-cancer patients. The CCP-CANCER UK will provide valuable information that would educate as well as help inform current practice and development of guidelines globally with regard to COVID19 infection in cancer patients. While samples collected within CCP-UK from cancer patients will enable an understanding of the biology of COVID-19 in the setting of cancer-related immunodeficiency both innate and iatrogenic.

ELIGIBILITY:
Inclusion Criteria:

- Patients with proven COVID-19 and a diagnosis of cancer who are enrolled into any Tier of the Principal CCP-UK protocol.

Exclusion Criteria:

- None in addition to those specified in the Principal CCP-UK protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are enrolled on to the CCP UK protocol study with COVID-19 and subsequently determined to have a concurrent or history of cancer
Sampling Method: Probability Sample
Enrollment: 9000 (Actual)
Dates: Start 2021-02-28 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
To determine the COVID-19 fatality rate overall in the cancer population using the most up to date dataset from the first wave. | 12 months
  Death rate among cohort of cancer and COVID-19 patients
To determine the COVID-19 fatality rate in different tumour types. | 12 months
  Exploring the number of deaths per group when sub grouping tumour types

SECONDARY OUTCOMES:
To describe the clinical features and severity of COVID-19 in different tumour types. | 12 months
  Comparison of the outcomes in COVID-19 across various tumour groups
To identify other clinical and laboratory variables that correlate with COVID-19 severity and mortality in different tumour types. | 12 months
  The rate of death and outcomes in COVID-19 will be subgrouped across various tumour types and compared against various clinical and laboratory indicators from the dataset and translational analysis
To determine the influence of disease stage, treatment intent and treatment history on severity and COVID-19 fatality rate. | 12 months
  Trends in stage of cancer at COVID-19 diagnosis, the treatment modalities administered both concurrently and previously will be compared against poorer outcomes and sequela for trends. Severity and Frailty with be stratified across all 3 factors, this is one outcome.
To describe the use of healthcare resources (including intensive care) in the treatment of COVID-19 in different tumour types. | 12 months
  To compare the admission time, interventions and assessments needed for the treatment of COVID-19 across various Tumour types. For each tumour type, the admission, intervention and assessments will be collated and compared with other tumour types. This is one outcome.
To undertake a matched cohort study using the cancer and non-cancer patients with COVID-19. | 12 months
  The Cancer Data set will be linked with the main CCP UK study for an overall comparison in COVID-19 outcomes and interventions in patient who have cancer and those who do not have cancer

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Palmieri, Principal Investigator — Clatterbridge Cancer Centre NHS Foundation Trust; Lance Turtle, Principal Investigator — University of Liverpool
Locations (1):
- The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The Cancer cohort data is being shared with the University of Edinburgh, within their data safe haven, in order to link with main cohort data. The UoE safe haven is part of the CCP Cancer study and not external researchers.